CLINICAL TRIAL: NCT01340118
Title: Concurrent Improvement of Exhaled Nitric Oxide and FEF25-75 After Treatment With Inhaled Corticosteroid in Children With Controlled Asthma
Brief Title: Improvement of FeNO and FEF25-75 After Inhaled Corticosteroid Treatment of Asthma
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chungbuk National University (Other)
Responsible Party: Youn-soo hahn, Department of pediatics,Department of Pediatrics, College of Medicine and Medical Research Institute, Chungbuk National University, Cheongju, Korea,
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WC asthma treatment based FeNO
Record Dates: First submitted 2011-04-15; First posted 2011-04-22 (Estimated); Last update posted 2011-04-22 (Estimated); Status verified 2011-04

CONDITIONS: Asthma
Keywords: Asthma; FEF25-75; exhaled nitric oxide; inhaled corticosteroid; children
MeSH Terms: conditions — Asthma | interventions — Budesonide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Budesonide (Experimental): Patients with FeNO level greater than 25 ppb were randomly allocated to one of two groups. Randomisation was stratified by baseline FeNO. In one group (treatment group), participants were assigned to once daily treatment with 400 µg budesonide. In the other group (non-treatment group), participants did not receive any medication.
  Interventions: Drug: Budesonide
- remain untreated (No Intervention)

INTERVENTIONS:
Drug: Budesonide — once daily inhalation with 400 µg budesonide (dry powder)during 6 weeks
  Arms: Budesonide

SUMMARY:
Abnormal lung function and high exhaled nitric oxide (FeNO) have been reported in asymptomatic patients with asthma. The investigators aimed to assess whether FeNO and FEF25-75 improve concurrently after treatment with inhaled corticosteroid (ICS) in patients with controlled asthma. Geometric mean (GM) FeNO and spirometric values in patients 8 to 16 years of age who maintained asthma control without controller medication were compared with healthy controls and patients with uncontrolled asthma who were also not receiving controller medications. Patients with controlled asthma and high FeNO (> 25 ppb) were randomized to ICS treatment or to remain untreated. Changes in spirometric values and GM FeNO from baseline were evaluated after 6 weeks.

DETAILED DESCRIPTION:
Current guideline-defined asthma control cannot be applied to the level of airway inflammation because neither symptoms nor the results of basic pulmonary function tests can reflect ongoing airway inflammation.Consequently, asymptomatic or minimally symptomatic patients are usually considered to have controlled asthma even if they have subclinical airway inflammation. Measures of airway inflammation are thus required to identify patients with silent airway inflammation which does not manifest itself as symptoms or impaired lung function. In addition, measurement should be easy to perform, reproducible, and associated with a high degree of acceptance by patients. In this regard, the advent of FeNO measurements represents a significant advance in monitoring airway inflammation of asthmatic patients. High FeNO values above certain cut-point may indicate active eosinophilic airway inflammation and the likelihood of deterioration in asthma control. However, it is still unclear that high FeNO in asymptomatic patients implies the need for the anti-inflammatory treatment.

Current guidelines for asthma management recommended forced expiratory volume in the first second (FEV1) as a principle spirometric parameter to assess airflow limitation. However, asthmatic subjects have air trapping in the presence of normal FEV1. Air trapping in asthmatic subjects has been demonstrated to be better correlated with forced expiratory flow between 25% and 75% of vital capacity % predicted (FEF25-75 % predicted) than FEV1 % predicted. In fact, impaired FEF25-75 is one of the most common abnormalities in pulmonary function in cross-sectional studies in asymptomatic patients. In addition, high FeNO in asymptomatic or minimally symptomatic patients may be accompanied by impairment of FEF25-75 because both parameters have been suggested to be measures of residual small airway disease. Therefore, there is a possibility that the improvement of FEF25-75 happens concomitantly with the decrease of FeNO during the anti-inflammatory treatment. In this study, we recruited previously well-documented atopic asthmatic children who required no medication to maintain asthma control for more than 3 months and had high FeNO levels (> 25 ppb). We aimed to assess whether the decrease of FeNO occurs simultaneously with improvement of FEF25-75 after treatment with inhaled corticosteroid (ICS) in these patients.

ELIGIBILITY:
Inclusion Criteria:

* sensitized to aeroallergens and previously diagnosed to have asthma based on the documentation of airway hyperresponsiveness (methacholine PC20 ≤ 8 mg/mL) and/or reversible airflow obstruction (≥ 12% improvement in FEV1 in response to inhaled beta 2-agonist)
* maintained asthma control without controller medication for 3 months or more
* FeNO > 25 ppb

Exclusion Criteria:

* who had significant pulmonary disease other than asthma or a history of gastroesophageal reflux

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 93 (Actual)
Dates: Start 2010-05; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
FeNO | 6 weeks after enrollment
  FeNO was measured at week 6 in the treatment and non-treatment groups.

SECONDARY OUTCOMES:
Spirometric values(FEF25-75,FEV1,FEV1/FVC) | 6 weeks
  Spirometric values were evaluated at week 6 in the treatment and non-treatment groups.
Asthma control test scores | 6 weeks
  Asthma control test scores were evaluated at week 6 in the treatment and non-treatment groups.

CONTACTS AND LOCATIONS:
Overall Officials: Youn-Soo Hahn, MD, PhD, Principal Investigator — Department of Pediatrics, College of Medicine and Medical Research Institute, Chungbuk National University, Cheongju
Locations (1):
- Chungbuk National University Hospital, Cheongju-si, North Chungcheong, South Korea